CLINICAL TRIAL: NCT03401281
Title: Randomised Trial of Different Dietary Fat Sources on Blood Lipids and Other CVD Risk Factors in Health Men and Women
Brief Title: Trial of Different Dietary Fat Sources on Blood Lipids and Other CVD Risk Factors
Acronym: COCHEESE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Gunter G C Kuhnle, Associate Professor in Nutrition and Health, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: GK001
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Dietary Modification
MeSH Terms: interventions — Coconut Oil; Butter; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Fats will be embedded in processed cheese - extend of masking will be assessed in sensory study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coconut oil (Active Comparator): 50g extra virgin coconut oil to be consumed daily for four weeks
  Interventions: Other: Coconut oil
- Butter (Active Comparator): 50g Butter to be consumed daily for four weeks
  Interventions: Other: Butter
- Olive oil (Active Comparator): 50g extra virgin olive oil to be consumed daily for four weeks
  Interventions: Other: Olive oil

INTERVENTIONS:
Other: Coconut oil — 50g extra virgin coconut oil daily for four weeks
  Arms: Coconut oil
Other: Butter — 50g butter daily for four weeks
  Arms: Butter
Other: Olive oil — 50g extra virgin olive oil daily for four weeks
  Arms: Olive oil

SUMMARY:
This is a randomised trial in which healthy volunteers, men and women aged 50-75 years from the general community are randomized into one of three arms: participants will be provided with 50 gm extra virgin coconut oil, or 50 grams butter or 50 extra virgin olive oil to be eaten daily for a month. The food will be provided in the form of processed cheese to mask participants. The key outcome is blood low density lipoprotein cholesterol concentrations and secondary outcomes blood lipid profile (total cholesterol, high density lipoprotein cholesterol, triglycerides) and anthropometric measures: weight and waist circumference. This trial is powered to detect a difference of 0.5 mmol/L LDL-cholesterol difference between the trial arms.

DETAILED DESCRIPTION:
This is a randomized trial in which healthy volunteers from the general community are randomized into one of three arms: consumption of 50 gm of extra virgin coconut oil daily OR 50gm of butter daily OR 50gm of extra virgin olive oil daily (50gm is about 2 ounces, or 2 table spoons), to be consumed over a one month period. The food will be provided in the form of processed cheese to mask participants.

After full informed consent, participants will attend an assessment visit and have a baseline measures of weight, height, waist circumference, blood pressure, a blood sample for assessment of blood lipids and other metabolic markers, and fill in a health questionnaire and dietary questionnaire. Participants will be randomly allocated to one of three arms: coconut oil, butter or olive oil and will be given supplies of these

After one month, participants will return for follow up assessment which will include a repeat blood sample, anthropometric measures and blood pressure, and questionnaire.

Blood samples collected by venipuncture will be stored at the University of Reading.

At the end of the study, all participants will be given the individual participant results of the anthropometric measures and lipid profiles at baseline and follow up as well as the overall findings of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the trial of dietary interventions for one month within the age range

Exclusion Criteria:

* No known cardiovascular disease: heart disease or stroke; no known cancer; no known diabetes; no use of lipid lowering medication eg. statins; no contraindications to high fat diet e.g. gall bladder or other gastrointestinal condition

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
LDL-Cholesterol | 4 weeks
  Blood LDL cholesterol concentrations

SECONDARY OUTCOMES:
Triglycerides | 4 weeks
  Blood triglycerides
HDL cholesterol | 4 weeks
  Blood HDL cholesterol
Total Cholesterol | 4 weeks
  Total Blood Cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, Please Select, United Kingdom

IPD SHARING:
Plan to Share IPD: No